CLINICAL TRIAL: NCT00622167
Title: Comparison of Dual Source Computed Tomography (DSCT) With Integrated Backscatter Intravascular Ultrasound (IB-IVUS) and Contrast Angiography in the Assessment of Coronary Artery Disease
Brief Title: Comparison of DSCT With IB-IVUS and Angiography in the Assessment of Coronary Artery Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment was slow, so enrollment has been closed.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007P001842
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: Plaque characteristics; DSCT; IVUS
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): All patients will receive integrated backscatter IVUS and dual source CT.
  Interventions: Device: Integrated Backscatter IVUS; Device: Dual Source Computed Tomography

INTERVENTIONS:
Device: Integrated Backscatter IVUS — All subjects have Integrated Backscatter IVUS and Dual Source CT imaging.
Device: Dual Source Computed Tomography — All subjects have DSCT and IBIVUS imaging

SUMMARY:
The purpose of this study is to compare different methods of looking at atherosclerotic plaques in heart arteries. Identifying the characteristics of these plaques noninvasively would be very valuable. This study is looking at a new CT scanner (DSCT) to noninvasively image these plaques compared to invasive ultrasound (the current standard).

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. To compare with contrast angiography, the ability of DSCT to detect and quantify coronary artery stenoses.
2. To compare with gray-scale IVUS, the ability of DSCT to quantify plaque cross-sectional diameter & area measurements & plaque volume.
3. To evaluate the ability of DSCT to assess plaque morphology and quantify plaque components as compared to gray-scale and IB-IVUS.
4. To evaluate the ability of DSCT to identify & measure lesion remodeling compared to gray-scale IVUS.
5. To determine if pre-PCI evaluation of coronary plaque morphology by IB-IVUS can a) predict procedural success as assessed by adequate stent strut apposition and expansion and b) peri-procedural myocardial necrosis as measured by biomarker elevation.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females
* > / = 18 years of age
* Scheduled for coronary angiography

Exclusion Criteria:

* Acute ST-elevation myocardial infarction within last 72 hours
* Current congestive heart failure
* Current cardiogenic shock
* Unstable clinical condition
* Known cardiomyopathy (EF < 30%)
* Creatinine >1.5 mg/dL
* Definite allergy to iodinated contrast media
* Current participation in an investigational drug or device research study
* HR > 65 and contraindications to the administration of beta blockers

Exclusion criteria assessed during catheterization procedure

* PCI of native coronary vessel not performed
* Left main stenosis > 50%
* Any vessel contraindicated for IVUS imaging
* Any lesion contraindicated for IVUS imaging
* Inability to pass IVUS catheter
* PCI of bifurcation lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from January 2008 until September 2008. The study ended early due to slow enrollment.
Pre-assignment Details: Subjects were consented prior to cardiac catheterization, and if they did not meet angiographic inclusion criteria they were withdrawn from the study.
Groups:
- IBIVUS and DSCT: All patients will receive integrated backscatter IVUS and dual source CT.
Period: Overall Study
Arm/Group | IBIVUS and DSCT
Started | 24
Completed | 4
Not Completed | 20
Not completed — Did not meet angiographic criteria | 20

BASELINE CHARACTERISTICS:
Arm/Group | IBIVUS and DSCT
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Study terminated after imaging 4 subjects due to slow enrollment. No analysis performed.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Plaque Characteristics Between DSCT (Dual Source Computed Tomography) and IVUS (Intravascular Ultrasound).
Description: Characteristics include plaque cross-sectional diameter, area measurements, plaque volume, and plaque morphology (composition).
Time Frame: At time of imaging
Population: Imaging 30 subjects was predicted to include enough plaques for analysis.
Measure: Number; unit: plaques
Units Other Than Participants: Plaques
Groups:
- Plaque Characteristics: Characteristics include plaque cross-sectional diameter, area measurements, plaque volume, and plaque morphology.
Arm/Group | Plaque Characteristics
Number analyzed (Participants) | 0
Number analyzed (Plaques) | 0
Statistical Analysis 1: Comparison: Plaque Characteristics; Plaque characteristics including plaque cross-sectional diameter, area measurements, plaque volume, and plaque morphology would be compared between IBIVUS, DSCT and angiography; Test type: Superiority or Other; p = 0, Not done

ADVERSE EVENTS:
Description: Total number of subjects at risk=4 since 20 subjects were screen failures and did not have any study imaging.
Arm/Group | IBIVUS and DSCT
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Study terminated after imaging 4 subjects due to slow enrollment. Results will not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes